CLINICAL TRIAL: NCT03246451
Title: The Role of GLP-1 Receptor Signalling in the Glucose-lowering Effect of Metformin During Meal Ingestion in Patients With T2D
Brief Title: The Role of GLP-1 Receptor Signalling in the Glucose-lowering Effect of Metformin in Patients With T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Laura Smidt Hansen, Bachelor of Science, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UHG-CFD-METEX
Record Dates: First submitted 2017-08-01; First posted 2017-08-11 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Glucose Metabolism Disorders
Keywords: GLP-1; glucagon-like peptide-1; Metformin; Exendin(9-39)
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Metformin; Sodium Chloride; exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo, oral tablet in 14 days and in liquid meal.
  Interventions: Drug: Placebo Oral Tablet
- Metformin (Experimental): Metformin, oral tablet 2-4 x 500 mg in 14 days and in liquid meal.
  Interventions: Drug: Metformin
- Saline (Experimental): Saline infusion (9mg/mL) on experimental days
  Interventions: Drug: Saline
- Exendin(9-39) (Experimental): Exendin(9-39) infusion. GLP-1 receptor antagonist used as a study tool on experimental days.
  Interventions: Drug: Exendin (9-39)

INTERVENTIONS:
Drug: Placebo Oral Tablet — 2-4 tablets in 14 days
  Arms: Placebo
Drug: Metformin — 1000-2000 mg in 14 days
  Arms: Metformin
Drug: Saline — 9 mg/ml saline infusion during experimental days
  Arms: Saline
Drug: Exendin (9-39) — Infusion of GLP-1 receptor antagonist used as a tool during experimental days
  Arms: Exendin(9-39)

SUMMARY:
Delineation of the role of glucagon-like peptide-1 receptor signalling in the glucose-lowering effect of metformin during meal ingestion in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Aim: To evaluate the contribution of metformin-induced GLP-1 secretion on the glucose-lowering effect of metformin in patients with type 2 diabetes treated with metformin for 14 days. Furthermore, the investigators aim to elucidate the mechanisms by which metformin-induced GLP-1 secretion may affect glucose levels in patients with type 2 diabetes.

Fifteen patients with type 2 diabetes treated with lifestyle intervention and/or metformin as the only glucose-lowering drug will be enrolled in the study. The effect of a 14-day metformin treatment course on postprandial glucose tolerance will be examined with and without infusion of the GLP-1 receptor antagonist exendin9-39 in 15 patients with type 2 diabetes.

The double-blinded, placebo-controlled, randomised, cross-over study consists of four study days with concomitant infusions of A) placebo + placebo, B) placebo + exendin9-39, C) metformin + placebo and D) metformin + exendin9-39.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least three months (diagnosed according to the criteria of the World Health Organization (WHO)), with a HbA1c <58 mmol/mol.
* Caucasian ethnicity
* Lifestyle intervention and/or metformin monotherapy
* Normal haemoglobin
* Age >18 years
* BMI >23 kg/m2 and <35 kg/m2
* Informed and written consent

Exclusion Criteria:

* Liver disease
* Gastrointestinal disease, previous intestinal resection, cholecystectomy or any major intra-abdominal surgery
* Hypo- or hyperphosphataemia
* Reduced kidney function or nephropathy
* Treatment with medicine that cannot be paused for 12 hours
* Intake of antibiotics two months prior to study
* Hypo- or hypercalcaemia
* Hypo- and hyperthyroidism
* Treatment with oral anticoagulants
* Active or recent malignant disease
* Any treatment or condition requiring acute or sub-acute medical or surgical intervention
* Lack of effective birth control in premenopausal women
* Positive pregnancy test on study days in premenopausal women
* Pregnancy
* Women who are breastfeeding
* Any condition considered incompatible with participation by the investigators
* If the subjects receive any antibiotic treatment while included in the study they will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2017-12-10 (Actual)

PRIMARY OUTCOMES:
Plasma glucose | Minutes 240
  The difference between the effect of metformin on postprandial glucose tolerance (as assessed by area under curve (AUC) for plasma glucose during a standardised liquid mixed meal test) with and without blockade of GLP-1 signalling by exendin 9-39.

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Study Director — UHGentofte, Center for Diabetes Research
Locations (1):
- Center for Diabetes Research, Gentofte Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen LS, Gasbjerg LS, Bronden A, Dalsgaard NB, Bahne E, Stensen S, Hellmann PH, Rehfeld JF, Hartmann B, Wewer Albrechtsen NJ, Holst JJ, Vilsboll T, Knop FK. The role of glucagon-like peptide 1 in the postprandial effects of metformin in type 2 diabetes: a randomized crossover trial. Eur J Endocrinol. 2024 Aug 5;191(2):192-203. doi: 10.1093/ejendo/lvae095. PMID 39049802